CLINICAL TRIAL: NCT03688659
Title: Treatment of Infective Endocarditis by Vancomycin and Gentamycin in Assiut University Children Hospital
Brief Title: Vancomycin, Gentamycin in Infective Endocarditis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Sarah Sobhy Habib, principal investigator, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: vgie
Record Dates: First submitted 2018-09-19; First posted 2018-09-28 (Actual); Last update posted 2018-09-28 (Actual); Status verified 2018-09

CONDITIONS: Infective Endocarditis
MeSH Terms: conditions — Endocarditis | interventions — Vancomycin; Gentamicins

STUDY DESIGN:
Masking Description: open
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- vancomycin,gentamycin in endocarditis (Other): patients with infective endocarditis will recieve intravenous infusion Vancomycin 30 mg/kg/day for 4:6 weeks and intravenous Gentamycin 3mg/kg/day for 2 weeks
  Interventions: Drug: Vancomycin and gentamycin

INTERVENTIONS:
Drug: Vancomycin and gentamycin — intravenous
  Other Names: vancomycin and geramycin

SUMMARY:
Infective endocarditis is a microbial infection of the endocardial surface of the heart.

DETAILED DESCRIPTION:
Infective endocarditis is usually suspected in a patient with fever and a new or changing cardiac murmur and is diagnosed based on the presence of a vegetation on echocardiography and positive blood cultures. Diagnosis of endocarditis is usually easy in febrile patients with a continuous bacteremia and the presence of vegetation on echocardiography Infective endocarditis includes bacterial endocarditis ( streptococcus viridans, enterococci and staphylococcus aureus are the main causes), as well as non bacterial endocarditis as those caused by viruses, fungi, chlamydia and rickettsia. It is usually superimposed on underlying congenital or rheumatic cardiac lesions, it also could occur in patients who had central vwnous catheter without underlying cardiac abnormality.

Infective endocarditis has been clinically divided into acute and subacute presentation. Acute bacterial endocarditis is a fulminant illness over days to weeks (<2 weeks), and is more likely due to Staphylococcus aureus which has much greater virulence. Subacute bacterial endocarditis is often due to Streptococci of low virulence and mild to moderate illness which progresses slowly over weeks and months (>2 weeks).

Bacterial endocarditis is a disease in which complete eradication of the organism is required. Bacteria involved in endocarditis are relatively protected from phagocytic activity by the vegetation, which contains high concentrations of bacteria with relatively low metabolic rates. Prolonged parenteral therapy is the only way to achieve bactericidal serum levels for the time needed to kill all the bacteria present in a vegetation of endocarditis. Treatment generally ranges from 4-8 weeks.

Patient with native valve endocarditis caused by S.Pneumoniae may be given penicillin with or without aminoglycosides.

combining an antistaphylococcal penicillin with an aminoglycoside covers against S.viridan,S.aureus and grame_negative organisms.

vancomycin can be substituted for a semisynthetic penicillin if methecillin_resistant staphylococcus aureus infection or penicillin allergy is suspected vancomycin plus gentamycin for 4 weeks is recommended for those who are unable to tolerate B-lactam antibiotic agents,and is associated with faster clearing of bactereamia Investigation; positive blood culture leucocytosis elevated acute phase reactants like CRP, ESR anemia in long standing cases echocardiography Treatment hospitalization and bed rest treatment of heart failure using of anti coagulant therapy. antimicrobial agents:

* several general principles provide a basis for the treatment
* the choice of antimicrobial therapy depends on the organism and its sensetivity pattern
* parenteral therapy specially in infants and childern
* prolonged course usually 4-6weeks
* bactericidal agents
* synergetic combination: the usual initial regimens an antistaphlococcal semisynthetic penicillin and an aminoglycoside(Gentamycin),if a methicillin resistant S.aureus is suspected ,vancomycin should be substituted for the semisynthetic penicillin.

vancomycin should be used in place of penicillin or semisynthetic penicillin in penicillin allergic patients vancomycin should be used in cases with echocardiographic signs of infective endocarditis in addition to gentamycin Surgical intervention; surgical debridment of infected material and replacement of the valve with a mechanical or bioprosthetic artificial heart valve is necessary in certain situations.

* patients with significant valve stenosis or regurgitation causing heart failure.
* recurrent septic emboli despite appropriate antibiotic treatment
* large vegetation (> 10 mm)
* abscess formation
* early closure of mitral valve

ELIGIBILITY:
Inclusion Criteria:

1. patients with cardiac proplem having infective endocaditis.
2. patients are newly diagnosed as recent intracardiac vegetations .

Exclusion Criteria:

1.patients are old diagnosed as intracardiac vegetations more than 6 months

Ages: 1 Week to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-01-01 (Estimated); Primary Completion 2021-01-01 (Estimated); Study Completion 2021-01-01 (Estimated)

PRIMARY OUTCOMES:
vancomycin and gentamycin in infective endocarditis | 2 weeks
  using combination of intravenous vancomycin and intravenous gentamycin then assessment of patients by
  1. echocardiography to detect size of intracardiac vegetation

SECONDARY OUTCOMES:
vancomycin and gentamycin in infective endocarditis | 1 weeks
  using combination of intravenous vancomycin and intravenous gentamycin then assessment of patients by compelete blood picture to detect leucocytosis
vancomycin and gentamycin in infective endocarditis | 4 weeks
  using combination of intravenous vancomycin and intravenous gentamycin then assessment of patients by CRP if >6 means positive results